CLINICAL TRIAL: NCT00251004
Title: Efficacy and Safety Study Comparing Concentration-controlled Everolimus in Two Doses (1.5 and 3.0 mg/Day Starting Doses) With Reduced Cyclosporine Versus 1.44 g Mycophenolic Acid (as Sodium Salt) With Standard Dose Cyclosporine in de Novo Renal Transplant Recipients
Brief Title: Efficacy and Safety Study of Everolimus Plus Reduced Cyclosporine Versus Mycophenolic Acid Plus Cyclosporine in Kidney Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001A2309
Record Dates: First submitted 2005-11-07; First posted 2005-11-09 (Estimated); Results first posted 2011-05-10 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-04

CONDITIONS: Kidney Transplantation; Graft Rejection
Keywords: Renal transplantation, kidney, and organ transplant; Renal transplant rejection
MeSH Terms: interventions — Everolimus; Mycophenolic Acid; Cyclosporine; Basiliximab; Adrenal Cortex Hormones

ARMS (3):
- Low-dose Everolimus Group (Experimental): 1.5 mg everolimus (one 0.75-mg tablet bis in diem/twice a day (bid)) + basiliximab + reduced-dose Cyclosporine A (CsA) ± corticosteroids.
  The CsA dose was adjusted to attain a trough (C0) value within the pre-specified target ranges: starting at the day 5 visit: 100-200 ng/mL, starting at the month 2 visit: 75-150 ng/mL, starting at the month 4 visit: 50-100 ng/mL and starting at the month 6 visit: 25-50 ng/mL. Patients received their first dose of basiliximab within 2 hours prior to transplant surgery and on day 4 post-transplant or according to local practice. Corticosteroids were administered according to local therapy.
  Interventions: Drug: Everolimus; Drug: Cyclosporine A (CsA); Drug: Basiliximab; Drug: Corticosteroids
- High-dose Everolimus Group (Experimental): 3.0 mg everolimus (two 0.75-mg tablets bid) + basiliximab + reduced-dose CsA ± corticosteroids.
  The CsA dose was adjusted to attain a trough (C0) value within the pre-specified target ranges: starting at the day 5 visit: 100-200 ng/mL, starting at the month 2 visit: 75-150 ng/mL, starting at the month 4 visit: 50-100 ng/mL and starting at the month 6 visit: 25-50 ng/mL. Patients received their first dose of basiliximab within 2 hours prior to transplant surgery and on day 4 post-transplant or according to local practice. Corticosteroids were administered according to local therapy.
  Interventions: Drug: Everolimus; Drug: Cyclosporine A (CsA); Drug: Basiliximab; Drug: Corticosteroids
- Control Group (Active Comparator): 1.44 g Mycophenolic Acid (two 360-mg tablets bid) + basiliximab + standard-dose CsA ± corticosteroids.
  The CsA dose was adjusted to attain a C0 value within the following range for the time of the study: starting at the day 5 visit: 200-300 ng/mL, starting at the month 2 visit and thereafter: 100-250 ng/mL. Patients received their first dose of basiliximab within 2 hours prior to transplant surgery and on day 4 post-transplant or according to local practice. Corticosteroids were administered according to local therapy.
  Interventions: Drug: Mycophenolic Acid (MPA); Drug: Cyclosporine A (CsA); Drug: Basiliximab; Drug: Corticosteroids

INTERVENTIONS:
Drug: Everolimus — oral, bis in diem/twice a day (bid)
  Other Names: Certican, Zotress
  Arms: High-dose Everolimus Group; Low-dose Everolimus Group
Drug: Mycophenolic Acid (MPA) — 2 oral capsules of mycophenolic acid 360mg administered bid
  Other Names: Myfortic
  Arms: Control Group
Drug: Cyclosporine A (CsA) — CsA dose adjustments were based on CsA trough levels (C0).
  Other Names: Neoral
Drug: Basiliximab — All patients received two 20 mg doses of basiliximab administered intravenously. The first dose was to be given within 2 hours prior to transplant surgery and the second dose was to be administered on day 4, or each dose could have been administered according to local practice.
  Other Names: Simulect
Drug: Corticosteroids — Oral corticosteroids were administered according to local practice during the trial. At the same center, all patients were to follow the same steroid administration protocol.

SUMMARY:
The purpose of this study was to compare the safety and efficacy of three immunosuppressive treatment regimens following a kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of any race between 18 to 70 years old (inclusive)
* Patients who gave written informed consent to participate in the study

Exclusion Criteria:

* Recipients of multi-organ transplantation
* Recipients of a primary cadaveric or primary non-human leucocyte antigen (HLA) identical living donor kidney transplantation.
* Graft cold ischemia time greater than 40 hours.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 833 (Actual)
Dates: Start 2005-10; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Wajih Z, Karpe KM, Walters GD. Interventions for BK virus infection in kidney transplant recipients. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD013344. doi: 10.1002/14651858.CD013344.pub2. PMID 39382091
- [Derived] Cibrik D, Silva HT Jr, Vathsala A, Lackova E, Cornu-Artis C, Walker RG, Wang Z, Zibari GB, Shihab F, Kim YS. Randomized trial of everolimus-facilitated calcineurin inhibitor minimization over 24 months in renal transplantation. Transplantation. 2013 Apr 15;95(7):933-42. doi: 10.1097/TP.0b013e3182848e03. PMID 23422495
- [Derived] Shihab FS, Cibrik D, Chan L, Kim YS, Carmellini M, Walker R, Zibari G, Pattison J, Cornu-Artis C, Wang Z, Tedesco-Silva H Jr. Association of clinical events with everolimus exposure in kidney transplant patients receiving reduced cyclosporine. Clin Transplant. 2013 Mar-Apr;27(2):217-26. doi: 10.1111/ctr.12045. Epub 2012 Dec 12. PMID 23230975

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: 1.44 g Mycophenolic Acid (MPA) (two 360-mg tablets bid) + basiliximab + standard-dose CsA ± corticosteroids.
  The CsA dose was adjusted to attain a C0 value within the following range for the time of the study: starting at the day 5 visit: 200-300 ng/mL, starting at the month 2 visit and thereafter: 100-250 ng/mL. Patients received their first dose of basiliximab within 2 hours prior to transplant surgery and on day 4 post-transplant or according to local practice. Corticosteroids were administered according to local therapy.
Period: Overall Study
Arm/Group | Low-dose Everolimus Group | High-dose Everolimus Group | Control Group
Started | 277 | 279 | 277
12 Month Analysis | 241 (Under 12 month analysis under group 1, 179 Completed study medication.) | 249 (Under 12 month analysis under group 2, 175 Completed study medication.) | 253 (Under 12 month analysis under group 3, 200 Completed study medication.)
24 Month Analysis | 232 (Under 24 month analysis under group 1, 167 Completed study medication.) | 238 (Under 24 month analysis under group 2, 161 Completed study medication.) | 246 (Under 24 month analysis under group 3, 185 Completed study medication.)
Completed | 232 | 238 | 246
Not Completed | 45 | 41 | 31
Not completed — Withdrawal by Subject | 23 | 16 | 14
Not completed — Death | 9 | 10 | 8
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Graft Loss | 12 | 13 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose Everolimus Group | High-dose Everolimus Group | Control Group | Total
Number analyzed (Participants) | 277 | 279 | 277 | 833
Age Continuous [Mean (Standard Deviation); unit: Years] | 45.7 (12.72) | 45.3 (13.36) | 47.2 (12.74) | 46.1 (12.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 88 | 88 | 276
  Male | 177 | 191 | 189 | 557

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite Efficacy Endpoints - 12 Month Analysis
Description: The primary efficacy endpoint was the 12 month analysis of primary efficacy failure defined as a composite endpoint including treated biopsy proven acute rejection (BPAR), graft loss, death or loss to follow-up. A treated BPAR episode was defined as a biopsy graded IA, IB, IIA, IIB, or III that was treated with anti-rejection therapy. Graft loss was defined as the allograft was presumed to be lost on the day the patient started dialysis and was not able to subsequently be removed from dialysis as well as re-transplant.
Time Frame: 12 months
Population: Intention-to-treat (ITT) population
Measure: Number; unit: Participants
Arm/Group | Low-dose Everolimus Group | High-dose Everolimus Group | Control Group
Number analyzed (Participants) | 277 | 279 | 277
Participants
  Composite Endpoint (n) | 75 | 60 | 70
  --Death | 8 | 9 | 6
  --Graft Loss | 13 | 13 | 9
  --Treated BPAR | 48 | 38 | 50
  --Lost to follow up | 12 | 6 | 9

2. Secondary Outcome: Percentage of Participants With the Composite Incidence of Graft Loss, Death or Loss to Follow up at 12 Months Post-transplantation
Description: Graft loss was defined as graft loss (the allograft was presumed to be lost on the day the patient started dialysis and was not able to subsequently be removed from dialysis) and re-transplant.
  A loss to follow-up patient in the composite endpoint of graft loss, death or loss to follow-up (the main secondary efficacy endpoint) was a patient who did not experience graft loss or death from day 1 and whose last day of contact was prior to study day 316.
Time Frame: 12 months
Population: Intention-to-treat (ITT) population.
Measure: Number; unit: Percentage of participants
Arm/Group | Low-dose Everolimus Group | High-dose Everolimus Group | Control Group
Number analyzed (Participants) | 277 | 279 | 277
Percentage of participants | 11.6 | 9.7 | 9.4
Statistical Analysis 1: Comparison: Low-dose Everolimus Group vs Control Group; Everolimus is non-inferior to mycophenolic acid (MPA) if the upper limit of the 95% confidence interval for the difference in combined graft loss, death or loss to follow-up rates is <10%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was set at 10%; p = 0.001, Z-test — To control for multiple comparisons, the two-sided significance level was set at 0.025; Difference in percentage = 2.2, 95% CI 2-sided [-2.9 to 7.3]
Statistical Analysis 2: Comparison: High-dose Everolimus Group vs Control Group; Everolimus is non-inferior to MPA if the upper limit of the 95% confidence interval for the difference in combined graft loss, death or loss to follow-up rates is <10%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was set at 10%; p < 0.001, Z-test — To control for multiple comparisons, the two-sided significance level was set at 0.025; Difference in Percentage = 0.3, 95% CI 2-sided [-4.6 to 5.2]

3. Primary Outcome: Non-inferiority Analysis on Percentage of Participants With Composite Efficacy Endpoints
Description: The primary efficacy endpoint was the 12 month analysis of primary efficacy failure defined as a composite endpoint including treated biopsy proven acute rejection (BPAR), graft loss, death or loss to follow-up. In the definition of composite efficacy failure, loss to follow-up includes patients who did not experience treated BPAR, graft loss or death on or after day 1 and whose last day of contact was prior to day 316, the start day of the 12 month visit window.
Time Frame: 12 months
Population: Intention-to-treat population
Measure: Number; unit: Percentage of Participants
Arm/Group | Low-dose Everolimus Group | High-dose Everolimus Group | Control Group
Number analyzed (Participants) | 277 | 279 | 277
Percentage of Participants | 27.1 | 21.5 | 25.3
Statistical Analysis 1: Comparison: Low-dose Everolimus Group vs Control Group; Everolimus is non-inferior to mycophenolic acid (MPA) if the upper limit of the 95% confidence interval for the difference in percentage of participants composite efficacy failure is <10%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was set at 10%; p = 0.014, Z - test — To control for multiple comparisons, the two-sided significance level was set at 0.025; Difference in percentage = 1.8, 95% CI 2-sided [-5.5 to 9.1]
Statistical Analysis 2: Comparison: High-dose Everolimus Group vs Control Group; Everolimus is non-inferior to MPA if the upper limit of the 95% confidence interval for the difference in composite efficacy failure rates is <10%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was set at 10%; p < 0.001, Z-test — To control for multiple comparisons, the two-sided significance level was set at 0.025; Difference in percentage = -3.8, 95% CI 2-sided [-10.8 to 3.3]

4. Secondary Outcome: Non-inferiority Analysis of Renal Function, Calculated by Glomerular Filtration Rate (cGFR) Using Modification of Diet in Renal Disease (MDRD) Formula
Description: Modification of Diet in Renal Disease (MDRD) formula is:
  GFR [mL/min/1.73m^2] = 186.3*(C^-1.154)*(A^-0.203)*G*R where
  * C is the serum concentration of creatinine [mg/dL],
  * A is patient age at sample collection date [years],
  * G=0.742 when gender is female, otherwise G=1,
  * R=1.21 when race is black, otherwise R=1
Time Frame: at 12 months
Population: Intention to treat (ITT) population.
Measure: Number; unit: mL/min/1.73m^2
Arm/Group | Low-dose Everolimus Group | High-dose Everolimus Group | Control Group
Number analyzed (Participants) | 277 | 279 | 277
mL/min/1.73m^2 | 54.66 [lower limit -1.6] | 51.41 [lower limit -4.9] | 52.24
Statistical Analysis 1: Comparison: Low-dose Everolimus Group vs Control Group; The null hypothesis: the mean GFR of the everolimus arm is lower (worse) than that of the MPA arm by 8 mL/min/1.73m^2 or more; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was set at -8 mL/min/1.73m^2; p < 0.001, t-test, 2 sided — To control for multiple comparisons, the two-sided significance level was set at 0.025; Mean Difference (Net) = 2.42, 95% CI 2-sided [-1.6 to 6.5]
Statistical Analysis 2: Comparison: High-dose Everolimus Group vs Control Group; [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was set at -8 mL/min/1.73m^2; p < 0.001, t-test, 2 sided — To control for multiple comparisons, the two-sided significance level was set at 0.025; Mean Difference (Net) = -0.83, 95% CI 2-sided [-4.9 to 3.3]

ADVERSE EVENTS:
Time Frame: At 24 month
Description: Safety population
Arm/Group | Low-dose Everolimus Group | High-dose Everolimus Group | Control Group
Serious Adverse Events (participants affected / at risk) | 176/274 | 193/278 | 168/273
Other Adverse Events (participants affected / at risk) | 268/274 | 272/278 | 264/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low-dose Everolimus Group (N=274) | High-dose Everolimus Group (N=278) | Control Group (N=273)
Anaemia (Blood and lymphatic system disorders) | 2 | 8 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 2
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 4 | 0
Angina pectoris (Cardiac disorders) | 2 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 4
Atrial flutter (Cardiac disorders) | 1 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 2 | 3
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 3 | 2 | 2
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2 | 0
Cardiomegaly (Cardiac disorders) | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 3 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 6 | 2
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 2
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0
Hyperparathyroidism tertiary (Endocrine disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 1 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 2 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 4
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 7 | 7
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 2 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 4
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 1 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 3 | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Sclerosing encapsulating peritonitis (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 2
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 7 | 6
Asthenia (General disorders) | 1 | 1 | 0
Chills (General disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 1 | 1 | 0
Hernia obstructive (General disorders) | 0 | 2 | 0
Implant site effusion (General disorders) | 1 | 1 | 0
Influenza like illness (General disorders) | 2 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 3 | 2
Oedema peripheral (General disorders) | 1 | 7 | 1
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 12 | 16 | 13
Sudden death (General disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 2 | 2
Hepatic cyst (Hepatobiliary disorders) | 1 | 0 | 0
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 | 0 | 0
Kidney transplant rejection (Immune system disorders) | 5 | 3 | 7
Serum sickness (Immune system disorders) | 0 | 0 | 1
Transplant rejection (Immune system disorders) | 1 | 0 | 1
Abdominal sepsis (Infections and infestations) | 1 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 2 | 0 | 0
Abscess (Infections and infestations) | 0 | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0
Arteriovenous fistula site infection (Infections and infestations) | 0 | 1 | 0
Arteriovenous graft site infection (Infections and infestations) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0
BK virus infection (Infections and infestations) | 1 | 0 | 2
Bacteraemia (Infections and infestations) | 4 | 2 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 2 | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 5 | 5 | 2
Cellulitis orbital (Infections and infestations) | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0
Clostridial infection (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Coccidioidomycosis (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 11
Cytomegalovirus oesophagitis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 6 | 4 | 9
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 1
Graft infection (Infections and infestations) | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 0 | 2
Herpes simplex (Infections and infestations) | 2 | 0 | 2
Herpes virus infection (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 6 | 5
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 1
Incision site infection (Infections and infestations) | 0 | 4 | 1
Infected lymphocele (Infections and infestations) | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 1
Localised infection (Infections and infestations) | 1 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 1
Osteomyelitis (Infections and infestations) | 3 | 3 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0
Papilloma viral infection (Infections and infestations) | 0 | 0 | 1
Parvovirus infection (Infections and infestations) | 0 | 1 | 0
Perinephric abscess (Infections and infestations) | 1 | 1 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 0 | 3
Pneumonia (Infections and infestations) | 8 | 13 | 12
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1
Polyomavirus-associated nephropathy (Infections and infestations) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 3 | 3
Pulmonary mycosis (Infections and infestations) | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 5 | 6 | 3
Pyelonephritis acute (Infections and infestations) | 1 | 7 | 1
Renal abscess (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 5 | 6 | 6
Septic shock (Infections and infestations) | 2 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Stent related infection (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 2 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 6
Urinary tract infection (Infections and infestations) | 20 | 22 | 25
Urosepsis (Infections and infestations) | 4 | 2 | 3
Viral infection (Infections and infestations) | 3 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Vulvovaginitis (Infections and infestations) | 0 | 0 | 1
West Nile viral infection (Infections and infestations) | 0 | 0 | 1
Wound abscess (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 4 | 3 | 2
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0
Wound sepsis (Infections and infestations) | 1 | 0 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 9 | 5 | 7
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Incision site haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 5 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Perinephric collection (Injury, poisoning and procedural complications) | 2 | 4 | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 2 | 2 | 4
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 0 | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 3 | 5 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 | 0 | 1
Post procedural urine leak (Injury, poisoning and procedural complications) | 2 | 4 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 2 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Pubic rami fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Renal graft loss (Injury, poisoning and procedural complications) | 14 | 18 | 9
Renal haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Renal injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Renal lymphocele (Injury, poisoning and procedural complications) | 0 | 2 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 3 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 2 | 4 | 5
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Transplant failure (Injury, poisoning and procedural complications) | 1 | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Urinary anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 1
Urinary bladder rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 3 | 1
Wound secretion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatine increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 20 | 19 | 22
Blood phosphorus increased (Investigations) | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1
Blood pressure increased (Investigations) | 2 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0
Cardiac enzymes increased (Investigations) | 0 | 1 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 1
Haematocrit decreased (Investigations) | 1 | 0 | 0
Hormone level abnormal (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Urine output decreased (Investigations) | 2 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 5 | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 3 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 7 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 3 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 3 | 2
Malnutrition (Metabolism and nutrition disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 4
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Primitive neuroectodermal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 3
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anoxic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Convulsion (Nervous system disorders) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0
Neurodegenerative disorder (Nervous system disorders) | 0 | 0 | 1
Neuromyopathy (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1
Stupor (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 3
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 2 | 1
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 5 | 4 | 4
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 4 | 4 | 7
IgA nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 1 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Renal artery stenosis (Renal and urinary disorders) | 3 | 2 | 3
Renal artery thrombosis (Renal and urinary disorders) | 1 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 6 | 7 | 7
Renal impairment (Renal and urinary disorders) | 7 | 2 | 3
Renal necrosis (Renal and urinary disorders) | 0 | 0 | 3
Renal tubular atrophy (Renal and urinary disorders) | 0 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 1 | 4 | 3
Residual urine (Renal and urinary disorders) | 0 | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 2 | 1
Ureteral necrosis (Renal and urinary disorders) | 2 | 1 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 6
Ureteric stenosis (Renal and urinary disorders) | 2 | 1 | 0
Urethral disorder (Renal and urinary disorders) | 1 | 0 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
Urinary fistula (Renal and urinary disorders) | 1 | 3 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 2 | 1 | 1
Urinoma (Renal and urinary disorders) | 1 | 1 | 1
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 1 | 0
Adnexa uteri mass (Reproductive system and breast disorders) | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 2 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alveolar proteinosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 9 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1
Blood pressure inadequately controlled (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 6 | 3 | 4
Essential hypertension (Vascular disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 1 | 1
Haemorrhage (Vascular disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 2 | 3
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 4 | 2
Hypovolaemic shock (Vascular disorders) | 0 | 2 | 0
Iliac artery stenosis (Vascular disorders) | 0 | 0 | 1
Lymphocele (Vascular disorders) | 15 | 15 | 8
Lymphorrhoea (Vascular disorders) | 2 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 2 | 0
Steal syndrome (Vascular disorders) | 0 | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low-dose Everolimus Group (N=274) | High-dose Everolimus Group (N=278) | Control Group (N=273)
Anaemia (Blood and lymphatic system disorders) | 75 | 86 | 67
Leukopenia (Blood and lymphatic system disorders) | 6 | 6 | 30
Polycythaemia (Blood and lymphatic system disorders) | 14 | 14 | 12
Tachycardia (Cardiac disorders) | 16 | 7 | 9
Abdominal distension (Gastrointestinal disorders) | 22 | 17 | 23
Abdominal pain (Gastrointestinal disorders) | 38 | 26 | 43
Abdominal pain upper (Gastrointestinal disorders) | 11 | 16 | 35
Constipation (Gastrointestinal disorders) | 107 | 125 | 116
Diarrhoea (Gastrointestinal disorders) | 59 | 52 | 65
Dyspepsia (Gastrointestinal disorders) | 18 | 21 | 38
Flatulence (Gastrointestinal disorders) | 15 | 9 | 11
Mouth ulceration (Gastrointestinal disorders) | 10 | 17 | 6
Nausea (Gastrointestinal disorders) | 85 | 81 | 91
Vomiting (Gastrointestinal disorders) | 44 | 46 | 65
Asthenia (General disorders) | 8 | 7 | 15
Fatigue (General disorders) | 33 | 23 | 31
Oedema (General disorders) | 23 | 20 | 19
Oedema peripheral (General disorders) | 134 | 126 | 116
Pyrexia (General disorders) | 51 | 55 | 38
Herpes zoster (Infections and infestations) | 12 | 8 | 14
Nasopharyngitis (Infections and infestations) | 19 | 25 | 18
Sinusitis (Infections and infestations) | 14 | 19 | 11
Upper respiratory tract infection (Infections and infestations) | 52 | 48 | 60
Urinary tract infection (Infections and infestations) | 62 | 59 | 60
Complications of transplant surgery (Injury, poisoning and procedural complications) | 10 | 14 | 12
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 18 | 27 | 18
Incision site pain (Injury, poisoning and procedural complications) | 48 | 56 | 45
Perinephric collection (Injury, poisoning and procedural complications) | 21 | 7 | 7
Post procedural discharge (Injury, poisoning and procedural complications) | 16 | 9 | 13
Procedural pain (Injury, poisoning and procedural complications) | 45 | 35 | 44
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 14 | 10 | 16
Blood creatinine increased (Investigations) | 40 | 38 | 53
Urine output decreased (Investigations) | 14 | 8 | 11
Weight increased (Investigations) | 22 | 23 | 33
Dehydration (Metabolism and nutrition disorders) | 14 | 13 | 11
Diabetes mellitus (Metabolism and nutrition disorders) | 12 | 22 | 19
Dyslipidaemia (Metabolism and nutrition disorders) | 41 | 38 | 26
Fluid overload (Metabolism and nutrition disorders) | 19 | 17 | 18
Hypercholesterolaemia (Metabolism and nutrition disorders) | 49 | 51 | 35
Hyperglycaemia (Metabolism and nutrition disorders) | 37 | 39 | 38
Hyperkalaemia (Metabolism and nutrition disorders) | 51 | 57 | 46
Hyperlipidaemia (Metabolism and nutrition disorders) | 55 | 62 | 44
Hyperphosphataemia (Metabolism and nutrition disorders) | 9 | 6 | 14
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 14 | 15 | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 28 | 30 | 22
Hypoglycaemia (Metabolism and nutrition disorders) | 17 | 11 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 37 | 47 | 32
Hypomagnesaemia (Metabolism and nutrition disorders) | 38 | 39 | 43
Hypophosphataemia (Metabolism and nutrition disorders) | 38 | 44 | 36
Metabolic acidosis (Metabolism and nutrition disorders) | 15 | 16 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 39 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 20 | 31
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 15 | 24
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 4 | 11
Osteopenia (Musculoskeletal and connective tissue disorders) | 16 | 12 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 36 | 29 | 33
Dizziness (Nervous system disorders) | 19 | 20 | 18
Headache (Nervous system disorders) | 55 | 49 | 46
Paraesthesia (Nervous system disorders) | 9 | 8 | 16
Tremor (Nervous system disorders) | 24 | 23 | 38
Anxiety (Psychiatric disorders) | 27 | 18 | 19
Insomnia (Psychiatric disorders) | 51 | 52 | 46
Dysuria (Renal and urinary disorders) | 29 | 28 | 30
Haematuria (Renal and urinary disorders) | 34 | 23 | 33
Proteinuria (Renal and urinary disorders) | 31 | 37 | 22
Renal tubular necrosis (Renal and urinary disorders) | 16 | 15 | 10
Erectile dysfunction (Reproductive system and breast disorders) | 11 | 15 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 29 | 35
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 21 | 29
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 | 16 | 12
Acne (Skin and subcutaneous tissue disorders) | 32 | 42 | 25
Hirsutism (Skin and subcutaneous tissue disorders) | 8 | 11 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 18 | 16
Rash (Skin and subcutaneous tissue disorders) | 13 | 17 | 17
Hypertension (Vascular disorders) | 86 | 83 | 87
Hypotension (Vascular disorders) | 17 | 24 | 26
Lymphocele (Vascular disorders) | 9 | 20 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.